CLINICAL TRIAL: NCT06183632
Title: Lipid Characterisation of Plasma Microparticles in a Large Population of Healthy Donors
Acronym: MicroLipids
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: LELEU 2023
Record Dates: First submitted 2023-12-14; First posted 2023-12-27 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Healthy Donor
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy donor: All healthy volunteers are eligible to donate according to EFS criteria.
  Interventions: Biological: blood sampling

INTERVENTIONS:
Biological: blood sampling — 3 x 7mL EDTA blood tubes

SUMMARY:
Extracellular vesicles (EVs) are membrane structures containing numerous mediators categorised according to their size and mode of production. Among them, microparticles (MPs) are EVs between 100 nm and 1 μm in size that are produced by budding at the plasma membrane of different cell types following different mechanisms of cell activation or death. MPs include a large pool of bioactive molecules, such as lipids, proteins or nucleic acids. This makes them important mediators of intercellular communication, increasingly recognised for their role in various biological processes such as inflammation, coagulation, immune response and tumour progression. Their ability to transmit molecular signals between cells may have implications for disease pathogenesis and cellular interactions in pathological microenvironments. These MPs therefore appear to be an innovative biomarker, potentially useful in the early management of disease, both in terms of diagnosis and as a therapeutic target.

The main techniques used to analyse these MPs include flow cytometry, which enables surface markers to be quantified and determined, and electron microscopy, which provides a direct view of their morphology and structure. Molecular biology, such as the quantitative PCR technique, is also an approach used by several teams, notably to search for RNA or DNA fragments involved in various biological processes. However, few studies have focused on the lipid composition of these MPs. Since MPs are membrane vesicles, they are a major lipid reservoir. In addition, lipids represent a significant population of molecules with extensive properties, whether in inflammation, cell proliferation, energy metabolism, etc.

The aim of this project is to develop a reliable and robust method for analysing plasma MP concentration, phenotype and lipid composition in a population of healthy volunteers. These parameters will subsequently provide a comparator for studying MPs in populations of patients suffering from cardiovascular and/or inflammatory diseases.

ELIGIBILITY:
Inclusion Criteria:

* Person who has given his/her non-opposition
* All healthy volunteers are eligible to donate according to EFS criteria.

Exclusion Criteria:

* Person subject to a legal protection measure (curatorship, guardianship, etc)
* Pregnant, parturient or breast-feeding women
* Adults who are incapable or unable to give their consent
* Minors
* Person not eligible to donate according to EFS criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be identified by EFS staff at the time of their appointment for a platelet donation at the EFS - Maison du Don, Dijon.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
microparticle concentration, phenotyping and lipid composition in a population of healthy subjects. | Through study completion, an average of 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France